CLINICAL TRIAL: NCT02936089
Title: Risk Stratification-directed Therapy for Acute Myeloid Leukemia With t(8;21) /AML1-ETO-positive
Brief Title: Risk Stratification-directed Therapy for AML With t(8;21) /AML1-ETO+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-2017-168
Record Dates: First submitted 2016-10-11; First posted 2016-10-18 (Estimated); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Acute Myeloid Leukemia; Risk Stratification
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Drug Therapy

STUDY DESIGN:
Intervention Model Description: Patients with newly diagnosed AML1/ETO-positive AML took risk-directed stratification therapy based on c-KIT and ASXL1 mutations and measurable residual disease (MRD). low risk (LR) group (KIT-ASXL1- with main molecular response (MMR)) was recommended to chemotherapy (CT) or autologous hematopoietic stem cell transplantation (auto-HSCT). Intermediate risk (IR) group (KIT+/ASXL1+ with MMR) was suggested for auto-HSCT or HLA-matched HSCT. High risk (HR) group (KIT+ASXL1+ or without MMR) was treated with allogeneic (allo-) HSCT.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low risk group (Experimental): Patients with KIT-ASXL1- (non-mutation, NM) and acquiring main molecular response (MMR) after two cycles of consolidation.
  Interventions: Other: Consolidation with chemotherapy (CT) or autologous hematopoietic stem cell transplantation (auto-HSCT)
- Intermediate risk group (Experimental): Patients with KIT+/ASXL1+ (single mutation, 1M) and acquiring MMR after two cycles of consolidation.
  Interventions: Other: Consolidation with auto-HSCT or HLA-matched HSCT
- High risk group (Experimental): Patients with KIT+ASXL1+ (two mutations ,2M) or without acquiring MMR after two cycles of consolidation.
  Interventions: Other: allogeneic HSCT

INTERVENTIONS:
Other: Consolidation with chemotherapy (CT) or autologous hematopoietic stem cell transplantation (auto-HSCT) — For CT, patients were treated with high dose cytarabine (HDAC), cytarabine at a dosage of 1-3 g/m2 q12 h ×6 doses, for 4-6 cycles.
  For auto-HSCT, patients were treated with 3 cycles of HDAC and then bridged to auto-HSCT.
  Arms: Low risk group
Other: Consolidation with auto-HSCT or HLA-matched HSCT — For auto-HSCT, patients were treated with 3 cycles of HDAC and then bridged to auto-HSCT.
  For HLA-matched HSCT, patients were treated with 1-2 cycles of HDAC and then bridged to HLA-matched HSCT. HLA-matched donors were available in these patients.
  Arms: Intermediate risk group
Other: allogeneic HSCT — For allogeneic HSCT, patients were treated with 1-2 cycles of HDAC and then bridged to allogeneic HSCT, including HLA-matched and haploidentical transplantation.
  Arms: High risk group

SUMMARY:
Acute myeloid leukemia with t(8;21) /AML1-ETO-positive (AE AML) is a heterogeneous disease entailing different prognoses. There were significant differences in the therapeutic effect between different subgroups of AE AML. Therefore, risk stratification-directed therapy is very necessary for AE AML.

DETAILED DESCRIPTION:
Acute myeloid leukemia with t(8;21) /AML1-ETO-positive (AE AML) is a heterogeneous disease entailing different prognoses.There were significant differences in the therapeutic effect between different subgroups of AE AML. For example, patients with c-kit mutation had higher relapse rate and lower overall survival, compared with those without c-kit mutation. Therefore, risk stratification-directed therapy is very necessary for AE AML. The purpose of this study is to establish risk stratification-directed therapy for AE AML.

ELIGIBILITY:
Inclusion Criteria:

* AE AML aged 14-70
* No abnormality in a vital sign (e.g., heart rate, respiratory rate, or blood pressure)
* Expected survival time is more than 2 months

Exclusion Criteria:

* Any abnormality in a vital sign (e.g., heart rate, respiratory rate, or blood pressure)
* Patients with any conditions not suitable for the trial (investigators' decision)

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2016-10; Primary Completion 2021-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
overall survival (OS) | 3 year

SECONDARY OUTCOMES:
leukemia relapse rate | 3 year
disease-free survival (DFS) | 3 year
event Free Survival (EFS) | 3 year

CONTACTS AND LOCATIONS:
Overall Officials: Dan Xu, Principal Investigator — Nanfang Hospital, Southern Medical University

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD, all IPD that underlie results will be shared in a publication. For the detail, those who are interested in can contact the authors.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will be available after being published, for at least five years.
Access Criteria: All collected IPD, all IPD that underlie results will be shared in a publication. For the detail, those who are interested in can contact the authors.

REFERENCES:
- [Derived] Xu D, Yang Y, Yin Z, Tu S, Nie D, Li Y, Huang Z, Sun Q, Huang C, Nie X, Yao Z, Shi P, Zhang Y, Jiang X, Liu Q, Yu G. Risk-directed therapy based on genetics and MRD improves the outcomes of AML1-ETO-positive AML patients, a multi-center prospective cohort study. Blood Cancer J. 2023 Nov 13;13(1):168. doi: 10.1038/s41408-023-00941-4. No abstract available. PMID 37957175